CLINICAL TRIAL: NCT00136448
Title: High-Dose Ara-C Followed by Continuous Infusion Interleukin-2 for Acute Myelogenous Leukemia in First Remission
Brief Title: High Dose Ara-C (HDAC) and Interleukin-2 (IL-2) for Patients With Acute Myelogenous Leukemia (AML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 92-148
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2011-03-10 (Estimated); Status verified 2011-03

CONDITIONS: Acute Myelogenous Leukemia
Keywords: AML; acute myelogenous leukemia; cytarabine; interleukin-2
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; Daunorubicin; Interleukin-2

INTERVENTIONS:
Drug: cytosine arabinoside (ara-C)
Drug: daunomycin
Drug: interleukin-2

SUMMARY:
This study will add interleukin-2 (IL-2) to a regimen of post-remission therapy consisting of high-dose ara-C. Patients with AML in first remission will receive 3 cycles of high-dose ara-C followed by continuous infusion and bolus interleukin-2 (IL-2). We, the researchers at the Dana-Farber Cancer Institute, plan to evaluate the immunologic effects of such treatment in these patients.

DETAILED DESCRIPTION:
Patients will receive standard remission induction therapy with daunorubicin at a dose of 45 mg/m2/day for 3 days and continuous infusion cytarabine at a dose of 200 mg/m2/day for 7 days.

Those patients who enter a remission status and have preserved liver and kidney function will then receive 3 cycles of post-remission therapy that will consist of high-dose cytarabine at a dose of 3000 mg/m2 every 12 (q12) hours on days 1, 3 and 5 (total of 6 doses).

Patients who are still in remission will receive interleukin-2 (IL-2) upon count recovery at a dose of 8.1 X 10^5 U/m2/day by continuous infusion for 10 weeks. In addition, patients will receive bolus IL-2 at a dose of 6 X 10^5 U/m2 by intravenous bolus weekly for 6 doses through day 63.

Patients will be seen on a weekly basis while on treatment for examination and bloodwork.

At the end of treatment, patients will have a physical exam and bloodwork performed monthly for two years, then 4 times per year for two years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have AML based on French-American-British (FAB) criteria.
* Patients must have a total bilirubin of < 2.0 mg/dL, SGOT < 90 IU/mL, alkaline phosphatase < 250 U/mL and a serum creatinine < 2.0 mg/dL.
* Age 18 years or greater.

Exclusion Criteria:

* History of an antecedent hematologic malignancy such as myelodysplastic syndromes (MDS).
* Uncontrolled infection.
* History of a previous or concomitant malignancy other than non-melanoma skin cancer.
* Evidence of central nervous system (CNS) leukemia.
* Current use of corticosteroids.
* Prior treatment for AML, other than hydroxyurea.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 1993-02; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The primary purpose of this study is to evaluate the ability of IL-2 to generate cytotoxic and inhibitory activity against cryopreserved autologous leukemic myeloblasts obtained at the time of diagnosis.

SECONDARY OUTCOMES:
To evaluate the safety of continuous infusion IL-2 with intermittent IL-2 boluses in patients with AML who have received 3 cycles of post-remission intensification therapy with high-dose ara-C
To assess additional immunologic effects of IL-2
To obtain preliminary data regarding the rate of disease relapse

CONTACTS AND LOCATIONS:
Overall Officials: Richard M. Stone, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States